CLINICAL TRIAL: NCT01716273
Title: A Randomised Controlled Trial to Investigate the Clinical and Cost-effectiveness of White Granulated Sugar Dressing Compared With Standard Treatment in the Management of Exudating Wounds With Parallel Economic Evaluation
Brief Title: Use of White Granulated Sugar on Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moses Murandu (Other)
Collaborators: Laboratoires URGO (Industry); University of Wolverhampton (Other); University of Birmingham (Other)
Responsible Party: Sponsor-Investigator, Moses Murandu, PhD student, University Hospital Birmingham
Organization: University Hospital Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRK4106
Record Dates: First submitted 2012-10-24; First posted 2012-10-29 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Infected Wounds
MeSH Terms: conditions — Wound Infection | interventions — Sucrose; Carboxymethylcellulose Sodium; sorbsan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic & Acute infected wounds (Experimental): Wound will be cleaned with normal saline or tap water and Granulated sugar will be applied directly to the wound and covered with an absorbent pad and held in place with a bandage and tape.
  Interventions: Other: Granulated Sugar; Other: Debridement Dressing
- Chronic and Acute infected wounds (Active Comparator): Wound will be cleaned with normal saline or tap water and an appropriate debridement dressing (Aquacel or Sorbsan) is applied to the wound and secured with a bandage and surgical tape.
  Interventions: Other: Granulated Sugar; Other: Debridement Dressing

INTERVENTIONS:
Other: Granulated Sugar — 30 grams of granulated sugar is used to cover the wound area and this is held in place using a dry dressing pad , bandage and tape.
  Other Names: Sucrose
Other: Debridement Dressing — 1 Aquacel or Sorbsan dressing will be put over the wound, and held in place with a dry dressing pad, bandage and tape.
  Other Names: Aquacel or Sorbsan

SUMMARY:
How effective is sugar in reducing the debriding of sloughy, necrotic or infected exudating wounds compared with standard treatment?

DETAILED DESCRIPTION:
Patients for whom all the following apply:

Have an exudating wound sizes 5cm2 and 40cm2 A minimum of 25% slough, infected and necrotic tissue No dry necrotic eschar present Ankle Brachial Pressure Index of greater than 0.6 Are over 18 years Independently and willingly consent

ELIGIBILITY:
Inclusion Criteria:

* Exudating wound sizes 5cm2 and 40cm2
* A minimum of 25% slough, infected and necrotic tissue
* No dry necrotic eschar
* Ankle Brachial Pressure Index of greater than 0.6
* Age over 18 years
* Able to independently and willingly consent

Exclusion Criteria:

* Participants in a trial evaluating other therapies for their wound
* Have previously been in this trial
* Women who are pregnant
* Participants not able to tolerate daily dressing change

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Time to debridement of wound | 4 weeks
  wounds will be photographed at entry into the study there after weekly till end of study at 4 weeks

SECONDARY OUTCOMES:
Reduction in wound surface area | 4 weeks
  Wound measurements will be taken at entry into the study then weekly until end of 4 weeks

OTHER OUTCOMES:
Quality of life | 4 weeks
  Participants will be given a QOL questionnaire to complete before commencing the treatment and at the end of the 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Simms, MBBSFRCS, Principal Investigator — University Hospital Birmingham NHS Fondation Trust; Moses Murandu, PhD student, Study Director — University of Wolverhampton
Locations (1):
- University Hospital Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Murandu M, Webber MA, Simms MH, Dealey C. Use of granulated sugar therapy in the management of sloughy or necrotic wounds: a pilot study. J Wound Care. 2011 May;20(5):206, 208, 210 passim. doi: 10.12968/jowc.2011.20.5.206. PMID 21647066